CLINICAL TRIAL: NCT03133429
Title: Badanie Kliniczne oceniające bezpieczeństwo i skuteczność Stosowania stentów Szyjnych MER® w Rewaskularyzacji tętnic Szyjnych.
Brief Title: Clinical Study to Evaluate the Safety and Effectiveness of MER® Stents in Carotid Revascularisation.
Acronym: MER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balton Sp.zo.o. (Industry)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MER
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Carotid Artery Stenosis
Keywords: carotid artery; stroke; stent
MeSH Terms: conditions — Carotid Stenosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with MER stent (Experimental): Patients eligible for Carotid Artery Stenting
  Interventions: Device: MER

INTERVENTIONS:
Device: MER — carotid artery stenting

SUMMARY:
The aim of the study is to confirm, whether the MER® stent can be used, without limitations, for the endovascular carotid stenosis treatment in daily clinical practice. Eligible patients will undergo the procedure of the common or internal carotid artery stenting using MER® with proximal or distal neuroprotection.

DETAILED DESCRIPTION:
MER® stent will be implanted in eligible patients with common and internal carotid stenosis after an informed consent.

Potential benefit of the MER® stent implantation will be evaluated based on angiography and duplex Doppler ultrasound examination.

Follow ups are scheduled at 30 days, 6 and 12 months after index procedure. Except for clinical follow up patients will undergo carotid vessels ultrasound examination after 6 and 12 months. In case of an emergency visit, caused by the Serious Adverse Event, Patient will undergo: neurological and cardiac evaluation as well as carotid vessels USG examination and extended CT or MRI scans.

In general, all procedures in the study will follow the local standard of care. The type of devices used during the angioplasty (including the MER® stents) will not differ from the devices used in the usual clinical practice in the hospital. DAPT and other medical therapy will be consistent with the rules of the Polish and European Society of Cardiology.

ELIGIBILITY:
Inclusion Criteria:

* De novo lesion located in the internal carotid artery or common carotid artery

  * DS ≥50% (nonsymptomatic patients) and ≤99% based on QCA
  * DS ≥75% (symptomatic patients) and ≤99% based on QCA
* Target lesion available for 20-60mm lenght and 4-10mm diameter scaffold
* Patient eligible for CAS
* Age ≥ 18
* Life expentancy ≥ 12 months
* The patient's written informed consent has been obtained prior to the procedure.

Exclusion Criteria:

* Lack of neurological CAS qualification
* The patient has experienced an acute myocardial infarction within 72 hours of the procedure
* The patient has known paroxysmal, persistent or permanent atrial fibrillation or flutter
* The patient has known gastrointestinal bleeding
* Pregnancy
* DAPT contraindications
* Surgery planned within 1 month after the procedure
* A platelet count <100,000/mm³ or >600,000/mm³
* The patient has known nickel, titanium or contrast allergy
* The target vessel is totally occluded
* The patient has stent(s) in the target lesion
* Statin therapy contraindications
* The target lesion has massive calcifications
* Hyperthyroidism
* Post-radiotherapy side effects
* No pulse in femoral artery
* Chronic kidney disease (creatinine level >2,0 mg/dl or eGFR<30 mL/min/1.73 m2 or dialysotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10; Primary Completion 2017-06-22 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Stroke within 30 days after the procedure | 30 days
  Stroke within 30 days after the procedure

SECONDARY OUTCOMES:
MAE | 30 days
  compound Major Adverse Events (death, stroke, heart attack) within 30 days after the procedure
MAE | 365 days
  compound Major Adverse Events (death, stroke, heart attack) within 365 days after the procedure. Restenosis (%DS ≥50%) within 365 days.
Target vessel revascularization within 365 days | 365 days
  Target vessel revascularization within 365 days
Procedure success | 365 days
  Procedure success (with residual stenosis ≤30%)
SADE | 365 days
  Serious Adverse Device Effect

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Odrowąż-Pieniążek, Prof., Principal Investigator — Oddział Kliniczny Chorób Serca i Naczyń Krakowski Szpital Specjalistyczny im. Jana Pawła II ul. Prądnicka 80 31-202 Kraków; Paweł Buszman, Prof., Principal Investigator — I Oddział Kardiologiczno-Angiologiczny American Heart of Poland S.A. ul. Sanatoryjna 1 43-450 Ustroń
Locations (4):
- Poland (4):
  - Małopolskie Centrum Sercowo-Naczyniowe PAKS American Heart of Poland S.A., Oddział Chirurgii naczyniowej, Chrzanów
  - Górnośląskie Centrum Medyczne im. prof. Leszka Gieca Uniwersytetu Medycznego w Katowicach, Oddział Chirurgii Ogólnej, Naczyń, Angiologii i Flebologii, Katowice
  - Oddział Kliniczny Chorób Serca i Naczyń Krakowski Szpital Specjalistyczny im. Jana Pawła II, Krakow
  - Centrum Interwencyjnego Leczenia Udaru i Chorób Naczyniowych Mózgu Instytut Psychiatrii i Neurologii, Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maciejewski D, Pieniazek P, Tekieli L, Paluszek P, Dzierwa K, Trystula M, Wojcik-Pedziwiatr M, Podolec P. Transradial approach for carotid artery stenting in a patient with severe peripheral arterial disease. Postepy Kardiol Interwencyjnej. 2014;10(1):47-9. doi: 10.5114/pwki.2014.41469. Epub 2014 Mar 23. PMID 24799929
- [Background] Dzierwa K, Pieniazek P, Tekieli L, Musialek P, Przewlocki T, Kablak-Ziembicka A, Kosobucka-Peszat R, Machnik R, Trystula M, Podolec P. Carotid artery stenting according to the "tailored CAS" algorithm performed in the very elderly patients: the thirty day outcome. Catheter Cardiovasc Interv. 2013 Nov 1;82(5):681-8. doi: 10.1002/ccd.25025. Epub 2013 Jul 3. PMID 23825008
- [Background] Pieniazek P, Tekieli L, Musialek P, Kablak Ziembicka A, Przewlocki T, Motyl R, Dzierwa K, Paluszek P, Hlawaty M, Zmudka K, Podolec P. Carotid artery stenting according to the tailored-CAS algorithm is associated with a low complication rate at 30 days: data from the TARGET-CAS study. Kardiol Pol. 2012;70(4):378-86. PMID 22528713
- [Background] Musialek P, Pieniazek P, Tracz W, Tekieli L, Przewlocki T, Kablak-Ziembicka A, Motyl R, Moczulski Z, Stepniewski J, Trystula M, Zajdel W, Roslawiecka A, Zmudka K, Podolec P. Safety of embolic protection device-assisted and unprotected intravascular ultrasound in evaluating carotid artery atherosclerotic lesions. Med Sci Monit. 2012 Feb;18(2):MT7-18. doi: 10.12659/msm.882452. PMID 22293887
- [Background] Dzierwa K, Pieniazek P, Musialek P, Piatek J, Tekieli L, Podolec P, Drwila R, Hlawaty M, Trystula M, Motyl R, Sadowski J. Treatment strategies in severe symptomatic carotid and coronary artery disease. Med Sci Monit. 2011 Aug;17(8):RA191-197. doi: 10.12659/msm.881896. PMID 21804476
- [Background] Pieniazek P. [A new era for the stenting of the carotid arteries in the light of the CREST study]. Kardiol Pol. 2010 Sep;68(9):1086-7. No abstract available. Polish. PMID 20859914